CLINICAL TRIAL: NCT02854540
Title: Management of Palmar Hyperhidrosis With Hydrogel-based Iontophoresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marlyanne Pol-Rodriguez, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37987
Record Dates: First submitted 2016-07-30; First posted 2016-08-03 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hyperhidrosis; Hyperhidrosis Palmaris et Plantaris
Keywords: hyperhidrosis; palmar; sweating; iontophoresis; sweat gland diseases; skin diseases
MeSH Terms: conditions — Hyperhidrosis; Hyperhidrosis Palmaris Et Plantaris; Sweat Gland Diseases; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hand A (iontophoresis) vs. Hand B (no treatment) (Experimental): During the treatment period, participants will be asked to treat one hand with the hydrogel electrode-based iontophoresis device. Participants will also be asked to leave the other hand untreated.
  Interventions: Device: Hydrogel electrode-based iontophoresis

INTERVENTIONS:
Device: Hydrogel electrode-based iontophoresis — Hydrogel was administered through iontophoresis, a process of transdermal drug delivery by use of a voltage gradient on the skin.

SUMMARY:
This study will evaluate the use of hydrogel electrode pads (rather than tap water baths) to deliver iontophoresis treatment using a traditional iontophoresis device. Participants will treat one hand with the hydrogel-based iontophoresis device and leave the other hand untreated.

DETAILED DESCRIPTION:
Palmar hyperhidrosis affects 4.3 million Americans and results in substantial quality of life impairment. Treatment options for palmar hyperhidrosis include antiperspirants, systemic anticholinergic agents, botulinum toxin injections, and iontophoresis. Standard iontophoresis involves submerging the hands in tap water through which current is applied to the palms for 30 minutes per day up to 3 times per week. While effective, treatment adherence rates are low.

This study will evaluate the use of hydrogel electrode pads (rather than tap water baths) to deliver iontophoresis treatment using a traditional iontophoresis device. Hydrogel electrode pads permit improved mobility and hand functionality during iontophoresis treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* 13 years of age or older
* >6 months self-reported history of primary palmar hyperhidrosis
* Initial gravimetry test: >20mg/min on each palm
* No topical treatments for hyperhidrosis (antiperspirants) on the palms for 2 weeks prior to the start of the study
* No systemic treatments for hyperhidrosis (anticholinergics) for 4 weeks prior to the start of the study
* No tap water iontophoresis treatment for 6 weeks
* No Botox injections on the palms for 6 months (if single treatment session) or 10 months (if >1 previous sessions) prior to the start of the study
* No history of cardiothoracic sympathectomy for hyperhidrosis
* Able to attend 3 office visits (Stanford Medical Outpatient Center located at 450 Broadway St, Redwood City, CA 94063; Lucile Packard Children's Hospital at 730 Welch Road, 1st Floor, Palo Alto, CA 94304) and one virtual visit in an 8 week time frame
* Capable of performing sweat level testing and hydrogel-based iontophoresis treatment at home, after training
* Hydrogel electrode pad fits on the hand (typically tip of middle finger to lower end of palm length of 6.5in (16.5cm) or greater)

Exclusion Criteria:

* Patients with implanted electronic medical devices e.g. pacemaker, implantable cardioverter/defibrillator)
* Patients with metal implants in the extremity that will be treated
* Patients with larger skin defects (on the palm or arm of the extremity that will be treated) that cannot be covered by petroleum jelly
* Pregnant or nursing women, or looking to become pregnant
* Patients on medications that interfere with neuroglandular transmission
* Patients with active infection locally or systemically
* Patients with history of contact dermatitis to acrylates
* Patients with history of contact or systemic allergy to iodine
* Patients with a history of ischemic heart disease, cardiac arrhythmias, epilepsy or thyroid disease

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlyanne Pol-Rodriguez, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Children's Health - Dermatology Department, Palo Alto, California
  - Stanford Medicine Outpatient Center, Redwood City, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MedlinePlus description of iontophoresis — https://medlineplus.gov/ency/article/007293.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Hand A was treated with hydrogel electrode-based iontophoresis. Hand B did not receive treatment.
  Hydrogel electrode-based iontophoresis: During the treatment period, participants were asked to treat one hand with the hydrogel electrode-based iontophoresis device. Participants were also asked to leave the other hand untreated.
Period: Overall Study
Arm/Group | All Participants
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Healthy teenagers and adults with a history of palmar hyperhidrosis
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Palmar Sweat Production
Description: Quantification of sweat production measured quantitatively using gravimetry, reported as milligrams of sweat per minute.
Time Frame: Baseline to week 2
Population: Two participants who were not able to tolerate the lower threshold dose were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mg/min
Units Other Than Participants: Hands
Groups:
- Hand A (Iontophoresis): Hand A was treated with hydrogel electrode-based iontophoresis.
  Hydrogel electrode-based iontophoresis: During the treatment period, participants were asked to treat one hand with the hydrogel electrode-based iontophoresis device. Participants were also asked to leave the other hand untreated.
- Hand B (no Treatment): Hand B did not receive treatment.
  Hydrogel electrode-based iontophoresis: During the treatment period, participants were asked to treat one hand with the hydrogel electrode-based iontophoresis device. Participants were also asked to leave the other hand untreated.
Arm/Group | Hand A (Iontophoresis) | Hand B (no Treatment)
Number analyzed (Participants) | 11 | 11
Number analyzed (Hands) | 11 | 11
mg/min
  Baseline | 44.8 (25.34) | 43.2 (24.77)
  Week 2 | 37.8 (41.07) | 24.9 (17.87)
Statistical Analysis 1: Comparison: Hand A (Iontophoresis) vs Hand B (no Treatment); Test type: Other; Mean difference (percent) = 59, Standard Deviation 16

2. Secondary Outcome: Patient Reported Pain (Visual Analogue Scale)
Description: Patient-reported pain on the treated hand using an 11-point visual analogue scale. Scale range: 0-10, with zero representing no pain, and 10 representing the worst pain imaginable.
  Participants recorded pain scores in a daily diary, and the score reported here is the average of all scores reported over the 2-week treatment period.
Time Frame: Baseline to week 2
Population: Two participants who were not able to tolerate the lower threshold dose were excluded from the analysis. This outcome was prespecified for the treated hand only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hand A (Iontophoresis)
Number analyzed (Participants) | 11
score on a scale | 1.7 (1.25)

3. Secondary Outcome: Modified Minor's Sweat Testing as a Quantitative Measure of Palmar Sweat Production
Description: Modified Minor's starch iodine testing, done with iodine imprints on plain paper, performed in office and at home to quantitatively measure sweat production.
Time Frame: Baseline to week 2
Population: No data were collected for this outcome measure.
Arm/Group | Hand A (Iontophoresis) | Hand B (no Treatment)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 week treatment period plus 6 week follow-up
Arm/Group | Hand A (Iontophoresis) | Hand B (no Treatment)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hand A (Iontophoresis) (N=13) | Hand B (no Treatment) (N=13)
itching (Skin and subcutaneous tissue disorders) | 6 | 0
blister (Skin and subcutaneous tissue disorders) | 2 | 0
crack/fissure (Skin and subcutaneous tissue disorders) | 1 | 0
minor skin burn (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT02854540/Prot_SAP_000.pdf